CLINICAL TRIAL: NCT00759603
Title: Lenalidomide in Combination With Rituximab as Treatment for Patients With Relapsed Chronic Lymphocytic Leukemia - RV-CLL-PI-0292
Brief Title: Lenalidomide and Rituximab as Treatment of Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0208; NCI-2012-01674 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Results first posted 2015-08-27 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-07

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: Leukemia; CLL; Chronic Lymphocytic Leukemia; SLL; Small Lymphocytic Lymphoma; Lenalidomide; Revlimid; Rituximab; Rituxan
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide + Rituximab (Experimental): Oral Lenalidomide 10 mg/day started on Day 9 of cycle 1; Rituximab 375 mg/m^2 intravenously on Day 1, Day 8, Day 15 and Day 22 then continued once every four weeks during cycles 3-12 (+ 7 days). Rituximab not given in Cycle 2. Treatment duration twelve cycles.
  Interventions: Drug: Lenalidomide; Drug: Rituximab

INTERVENTIONS:
Drug: Lenalidomide — Started on Day 9 of Cycle 1 at the dose of 10 mg/day and continued daily. Treatment duration will be twelve cycles.
  Other Names: Revlimid ®
Drug: Rituximab — Dose of 375 mg/m^2 given intravenously on Day 1, Day 8, Day 15 and Day 22 then continued once every four weeks during cycles 3-12 (+ 7 days). Rituximab not given in Cycle 2.
  Other Names: Rituxan®

SUMMARY:
The goal of this clinical research study is to learn if the combination of lenalidomide and rituximab can help to control Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL) in patients who have already received therapy. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Lenalidomide is designed to change the body's immune system and may also interfere with the development of tiny blood vessels that help support tumor growth. Therefore, in theory, it may decrease the growth of cancer cells.

Rituximab is designed to bind to a protein, called cluster of differentiation antigen 20 (CD20), that is on the surface of the leukemia cells, allowing the leukemia cells to be destroyed by the immune system.

Drug Administration:

If you are found to be eligible to take part in this study, you will receive rituximab through a needle into your vein 1 time a week in Cycle 1. You will not receive rituximab during Cycle 2, but you will continue to take lenalidomide.You will receive a dose of rituximab by vein on Day 1 of Cycles 3-12. Your first dose of rituximab will be given over 6-8 hours. If the first dose is well tolerated, you may receive the next doses over 2-4 hours. If the doctor thinks it is needed, the next doses may given over a longer time.

On Day 9 of Cycle 1, you will begin taking lenalidomide by mouth once a day. You will then take lenalidomide once a day, every day.

The dose and schedule of lenalidomide may change depending on the side effects you may experience. You should swallow lenalidomide capsules whole with a glass (8 ounces) water at the same time each day. Do not break, chew, or open the capsules. If you miss a dose of lenalidomide, take it as soon as you remember on the same day. If you miss a dose, it should NOT be made up on another day.

Each study cycle is 4 weeks.

Study Visits:

Once a week during the first 5 weeks, blood (about 1 tablespoon) will be drawn for routine tests.

After the first 5 weeks, blood (about 1 tablespoon) will be drawn for routine tests every 2 weeks until the doctor thinks your dose of lenalidomide will not change. After this, blood (about 1 tablespoon) will then be drawn every 4 weeks for routine tests.

At the end of Cycles 3, 6, and 12, you will have a bone marrow biopsy and aspirate to check the status of the disease. Blood (about 1 tablespoon) will be drawn for routine blood tests.

If you stay on study past 12 cycles, once every 6 cycles (Cycles 18, 24, 30, and so on), you will have a bone marrow biopsy and aspirate to check the status of the disease. Blood (about 1 tablespoon) will be drawn for routine blood tests.

Blood (about 1 tablespoon) will be drawn more often if the dose of lenalidomide needs to be changed or if you experience intolerable side effects.

Pregnancy Testing:

Women who are able to become pregnant must have a negative urine or blood (less than 1 teaspoon) pregnancy test 10-14 days and 24 hours before the first dose of lenalidomide, even if they have not had a menstrual period due to treatment of the disease or had only 1 menstrual period in the past 24 months.

If you have regular or no menstrual cycles, you will then have a urine or blood (less than 1 teaspoon) pregnancy test every week for the first 4 weeks, then every 4 weeks while taking lenalidomide, again as soon as you have been taken off of lenalidomide therapy, and then 28 days after you have stopped taking lenalidomide.

If you have irregular menstrual cycles, you will have urine or blood (less than 1 teaspoon) pregnancy test every week for the first 4 weeks, then every 2 weeks while taking lenalidomide, again as soon as you have been taken off of lenalidomide therapy, and then at 14 days and 28 days after you have stopped taking lenalidomide.

Length of Study:

You will be on study treatment for about 1 year. You will be taken off study early if you experience intolerable side effects or the disease gets worse.

If the doctor thinks you are benefiting, you may be able to continue taking the study treatment. If you continue, you will follow the same schedule of dosing and study visit schedule.

This is an investigational study. Lenalidomide and rituximab are FDA approved and commercially available. Lenalidomide is approved for the treatment of multiple myeloma and some myelodysplastic syndromes. Rituximab is approved for the treatment of chronic lymphoproliferative disorders and non-Hodgkin's lymphoma. The combination of these drugs to treat CLL and SLL is investigational.

Up to 60 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) with active disease.
2. Patients must be age 18 or over at the signing of consent and must understand and voluntarily sign an informed consent.
3. Prior treatment with purine analog based chemotherapy or chemoimmunotherapy.
4. Eastern Cooperative Oncology Group (ECOG)/World Health Organization (WHO) performance status of 0-2.
5. Adequate renal function indicated by serum creatinine less or equal to 2 mg/dl. Adequate hepatic function indicated as total bilirubin less or equal to 2 mg/dl and ALT less or equal to two times the upper limit of normal.
6. Disease free of prior malignancies for 3 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast. Patients with malignancies with indolent behavior such as prostate cancer treated with radiation or surgery can be enrolled in the study as long as they have a reasonable expectation to have been cured with the treatment modality received.
7. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test (sensitivity of at least 50 milli-International unit (mIU/mL) 10-14 days prior to starting lenalidomide. A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
8. Continued from Criteria #7. FCBP must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts talking lenalidomide. FCBP must also agree to ongoing pregnancy testing.
9. Continued from Criteria #8: Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
10. Men must agree not to father a child. They must agree to use a latex condom during sexual contact with females of childbearing potential while participating in the study and for at least 28 days following discontinuation from the study even if he has undergone a vasectomy. They will be warned that sharing study drug is prohibited and will be counseled about pregnancy precautions and potential risks of fetal exposure. They must agree to abstain from donating blood, semen, or sperm during study participation and for at least 28 days after discontinuation from the study.
11. Continued from Criteria #10: Counseling about the requirement for latex condom use during sexual contact with females of childbearing potential and the potential risks of fetal exposure must be conducted at a minimum of every 28 days. During counseling, subjects must be reminded not to share study drug and to not donate blood, sperm, or semen (during study participation and for 28 days following discontinuation from the study).

Exclusion Criteria:

1. Known sensitivity to lenalidomide or other thalidomide derivatives or rituximab.
2. Documented prolymphocytic leukemia (prolymphocytes more than 55% in the blood).
3. Known positivity for HIV or active hepatitis (B or C).
4. Pregnant or breast feeding females.
5. History of tuberculosis treated within the last five years or recent exposure to tuberculosis.
6. Any serious medical condition, laboratory abnormality, or psychiatric illness that places the subject at unacceptable risk if he/she were to participate in the study.
7. Patients with a recent history of deep vein thrombosis (DVT) or pulmonary embolus (PE), in the six months prior to enrollment are not eligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Ferrajoli, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Takahashi K, Hu B, Wang F, Yan Y, Kim E, Vitale C, Patel KP, Strati P, Gumbs C, Little L, Tippen S, Song X, Zhang J, Jain N, Thompson P, Garcia-Manero G, Kantarjian H, Estrov Z, Do KA, Keating M, Burger JA, Wierda WG, Futreal PA, Ferrajoli A. Clinical implications of cancer gene mutations in patients with chronic lymphocytic leukemia treated with lenalidomide. Blood. 2018 Apr 19;131(16):1820-1832. doi: 10.1182/blood-2017-11-817296. Epub 2018 Jan 22. PMID 29358183
- [Derived] Badoux XC, Keating MJ, Wen S, Wierda WG, O'Brien SM, Faderl S, Sargent R, Burger JA, Ferrajoli A. Phase II study of lenalidomide and rituximab as salvage therapy for patients with relapsed or refractory chronic lymphocytic leukemia. J Clin Oncol. 2013 Feb 10;31(5):584-91. doi: 10.1200/JCO.2012.42.8623. Epub 2012 Dec 26. PMID 23270003
- See also: University of Texas MD Anderson Cancer Center Website — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: September 22, 2008 to November 02, 2009. All recruitment done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: One of the 60 participants enrolled was excluded from the trial before any treatment assignment.
Period: Overall Study
Arm/Group | Lenalidomide + Rituximab
Started | 59
Completed | 59
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide + Rituximab
Number analyzed (Participants) | 59
Age, Continuous [Median (Full Range); unit: years] | 62 [42 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 46
Region of Enrollment [Number; unit: participants]
  United States | 59

OUTCOME MEASURES:

1. Primary Outcome: Overall Participant Response Rate: Percentage of Participants With Complete + Partial Response According to Revised National Cancer Institute-sponsored Working Group Guidelines
Description: Complete response: Absence lymphadenopathy, hepatomegaly or splenomegaly & constitutional symptoms; Normal complete blood count (CBC) exhibited by polymorphonuclear leukocytes>1500/µL, platelets>100,000/µL, hemoglobin>11.0 g/dL (untransfused); lymphocyte count <5,000/µL; Bone marrow aspirate & biopsy normocellular for age with <30% nucleated cells lymphocytes; Absence Lymphoid nodules. Fulfillment CR criteria after induction with exception of treatment related persistent cytopenia & bone marrow lymphoid nodules both considered partial response; Partial response: Requires 50% decrease in peripheral lymphocytes from pre-treatment, 50% reduction in lymphadenopathy, &/or 50% reduction in splenomegaly/hepatomegaly for 2+ months from therapy completion. Additionally one following from pre-treatment: Polymorphonuclear leukocytes 1,500/µL or 50% improvement; Platelets>100,000/µL or 50% improvement; Hemoglobin>11.0 g/dL (untransfused) or 50% improvement.
Time Frame: Responses assessed after 12 cycles, up to 48 weeks with interim assessments performed after 3, 6 and 12 cycles.
Measure: Number; unit: Percentage of Participants
Arm/Group | Lenalidomide + Rituximab
Number analyzed (Participants) | 59
Percentage of Participants | 66

ADVERSE EVENTS:
Time Frame: Adverse event collected through 12 cycles of 28-days.
Arm/Group | Lenalidomide + Rituximab
Serious Adverse Events (participants affected / at risk) | 29/59
Other Adverse Events (participants affected / at risk) | 59/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide + Rituximab (N=59)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 2 (3)
Cardiac arrhythmia (Cardiac disorders) | 1 (1)
Cardiac other (Cardiac disorders) | 1 (1)
Left ventricular diastolic dysfunction (Cardiac disorders) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Abdominal mass (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Abdominal pain (General disorders) | 1 (1)
Death (General disorders) | 2 (2)
Fever (General disorders) | 2 (3)
Tumor lysis syndrome (General disorders) | 1 (1)
Acute bronchitis (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Neutropenic fever (Infections and infestations) | 7 (8)
Perianal infection (Infections and infestations) | 1 (1)
Pulmonary infection RSV (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Syncope (Nervous system disorders) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 1 (1)
Elective surgery, right knee (Surgical and medical procedures) | 1 (1)
Autoimmune hemolytic anemia (Blood and lymphatic system disorders) | 1 (1)
Evan's syndrome (Blood and lymphatic system disorders) | 1 (1)
Left leg swelling (Blood and lymphatic system disorders) | 1 (1)
Thrombus (Cardiac disorders) | 1 (1)
Enteritis (Infections and infestations) | 2 (2)
Lung Infection (Infections and infestations) | 9 (17)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide + Rituximab (N=59)
Neutropenia (Blood and lymphatic system disorders) | 43 (43)
Thrombocytopenia (Blood and lymphatic system disorders) | 20 (20)
Anemia (Blood and lymphatic system disorders) | 9 (9)
Penumonia/bronchitis (Infections and infestations) | 6 (6)
fatigue (General disorders) | 32 (32)
Diarrhea (Gastrointestinal disorders) | 21 (21)
Tumor flare (General disorders) | 16 (16)
Sensory neuropathy (Nervous system disorders) | 14 (14)
Rash (Skin and subcutaneous tissue disorders) | 13 (13)
Constipation (Gastrointestinal disorders) | 11 (11)
Nausea (Gastrointestinal disorders) | 10 (10)
Neurologic other (Nervous system disorders) | 10 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (10)
Anorexia (Gastrointestinal disorders) | 9 (9)
Metabolic or laboratory (Metabolism and nutrition disorders) | 9 (9)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (8)
Elevated serum creatinine (Renal and urinary disorders) | 7 (7)
Gastrointestinal pain (General disorders) | 7 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 7 (7)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 7 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Peripheral edema (Blood and lymphatic system disorders) | 6 (6)
Heartburn (Gastrointestinal disorders) | 6 (6)
Headache (General disorders) | 6 (6)
Neutropenic fever (Infections and infestations) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes